CLINICAL TRIAL: NCT06707454
Title: Postoperative Clinical and Neurophysiological Assessment of Patients After Open Heart Surgery
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Osama Allam Ebrahim, Assistant Lecturer of Neuropsychiatry, Faculty of Medicine, Ain Shams University, Cairo, Egypt, Ain Shams University
Other Study IDs: FMASU MD115/2023
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Postoperative; Clinical; Neurophysiological Assessment; Open Heart Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients who will undergo open heart surgery, such as isolated coronary artery bypass grafting (CABG) or combined CABG and valve surgery.
  Interventions: Device: Digital Electroencephalography (DEEG)

INTERVENTIONS:
Device: Digital Electroencephalography (DEEG) — The enrolled patients will undergo Digital Electroencephalography (DEEG) monitoring for at least two hours. A senior epileptologist will make a DEEG interpretation to detect DEEG abnormality. DEEG patterns will be categorized according to the American Clinical Neurophysiology Society's standardized critical care DEEG terminology(normal, slowing and asymmetry, sharp and wave, periodic discharges, ictal patterns burst suppression, and electrocerebral silence)

SUMMARY:
This study aims to investigate postoperative clinical, cognitive and neurophysiological assessment of patients after open heart surgery among sample of Egyptian patients.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABAG) is one of the most common major surgical procedures, as more than 800,000 patients worldwide undergo myocardial revascularization procedures every year. Cardiopulmonary bypass (CPB) is an extracorporeal circulation procedure that assists the operation of cardiac and great vessels and is associated with perioperative morbidity and mortality.

Preoperative neurophysiological status as measured by electroencephalogram (EEG) had a specificity of 94.7% and a sensitivity of 76.9% for predicting 1-week postoperative cognitive status and with specificity of 78.3% and a sensitivity of 77.8% for predicting 3-months postoperative cognitive status.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 60 years.
* Both sexes.
* Patients who are scheduled for on-pump open heart surgery either isolated coronary artery bypass grafting (CABG) or combined CABG and valve surgery.

Exclusion Criteria:

* Patients with a past history of CNS disease (e.g. Epilepsy, brain tumors, or Dementia).
* Patients with metabolic disturbance.
* Illiterate patient.
* Patient with sever cognitive impairment on Mini-mental state Examination (MMSE) and/or Montreal Cognitive Assessment (MoCA)
* Patients who cannot undergo DEEG recordings (eg, uncooperative).
* Patients with abnormal brain images except for small vessel disease.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective observational study will be conducted on 80 patients undergoing pump open heart surgery, either isolated coronary artery bypass grafting (CABG) or combined CABG and valve surgery, at the Cardiothorathic Academy of Ain Shams University hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Neurological complications | 4 months postoperatively
  Neurological complications, including nonconvulsive seizures after open heart surgery, will be recorded.

SECONDARY OUTCOMES:
Electroencephalography (DEEG) monitoring | 24 hours postoperatively
  The enrolled patients will undergo Digital Electroencephalography (DEEG) monitoring for at least two hours. A senior epileptologist will interpret the DEEG to detect abnormalities. The DEEG patterns will be categorized according to the American Clinical Neurophysiology Society's standardized critical care DEEG terminology(normal, slowing and asymmetry, sharp and wave, periodic discharges, ictal patterns burst suppression, and electrocerebral silence).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.